CLINICAL TRIAL: NCT02415062
Title: The Efficacy of 23mg Versus 10mg of Donepezil in ParkInson's Disease With Dementia
Brief Title: The Efficacy and Safety Study of High Dose Donepezil in Parkinson's Disease With Dementia
Acronym: CUPID
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, Sangjin Kim, Busan Paik Hospital, Inje University, Inje University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CUPID-01
Record Dates: First submitted 2015-03-14; First posted 2015-04-14 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-08

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; dementia
MeSH Terms: conditions — Parkinson Disease; Dementia | interventions — Donepezil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- high dose donepezil (23mg) (Experimental): Patients with dementia in Parkinson's disease, who are treated with high dose donepezil (23mg)
  Interventions: Drug: Donepezil
- standard dose denepezil (10mg) (Active Comparator): Patients with dementia in Parkinson's disease, who are treated with standard dose donepezil (10mg)
  Interventions: Drug: Donepezil

INTERVENTIONS:
Drug: Donepezil — 23mg/day for 24 weeks versus 10mg/day for 24 weeks
  Other Names: aricept

SUMMARY:
The purpose of this study to evaluate the safety and efficacy of high-dose donepezil (23mg) in Parkinson's disease with dementia compared to standard dose donepezil.

DETAILED DESCRIPTION:
This study is open-label, prospective, randomized paralleled study. The investigators evaluate the efficacy of high-dose donepezil in patients with Parkinson's disease with dementia (PDD) who have taken standard donepezil (10mg) for 12 weeks. The participants, who sign the informed consent, are assigned into two groups randomly (high-dose donepezil group and standard donepezil group). All participants will be maintained the medication for 24 weeks and assessed cognitive function at 24 weeks. They will visit to clinic for 3 times (4, 12, 24 weeks) to assess cognitive function and adverse event. After the end of study, all participants were administrated by standard dose donepezil again.

ELIGIBILITY:
Inclusion criteria :

* Patients diagnosed as Parkinson's disease according to Queen Brain Bank criteria
* Patients who have been diagnosed as dementia after diagnosing Parkinson's disease at least 1 year.
* Patients with Hoehn and Yahr staging from 2 to 4
* Patients with MMSE score from 10 to 24
* Patients who have taken donepezil for at least 12 weeks before screening period
* Patients whose medications for Parkinson's disease have not change for 1 month
* Patients who give informed consent

Exclusion criteria :

* Patients who cannot be performed neuropsychiatric test because of hearing and visual difficulty
* Patients who have taken medicine affecting cognitive function such as anticholinergic drug and memantine -Patients diagnosed as dementia with Lewy body and vascular dementia-
* Patients who have history of neurosyphilis, head trauma, encephalitis or other movement disorders
* Patients who have psychiatric disease
* Except patients who are stable state under antidepressant or atypical neuroleptics
* Patients with child-bearing periods
* Patients who have severe liver or kidney disease necessary for aggressive treatment
* Patients who have gastrointestinal disease needed for treatment
* Patients who cannot taken tablet per oral
* Patients who are participated in other clinical trial except observational study

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Korean Mini-Mental State Examination-2 (MMSE-2) | 24 weeks
  scale for general cognitive function, We used Korean version of MMSE-2 from PAR company

SECONDARY OUTCOMES:
Korean-Instrumental Activities of Daily Living | 24 weeks
  scales for activities daily living
Clinical dementia rating | 24 weeks
  scales for activities of daily living
Unified Parkinson's disease rating scale (UPDRS) part 3 | 24 weeks
  scales for motor symptoms in Parkinson's disease
Modified Hoehn & Yahr stage | 24 weeks
  scales for status of Parkinson's disease
Schwab & England Activities of Daily Living | 24 weeks
  scales for activities daily living
Caregiver-Administered Neuropsychiatric Inventory | 24 weeks
  scales for status of caregiver
Global Deterioration Scale | 24 weeks
  scales for activities of daily living
Korean-Montreal Cognitive Assessment | 24 weeks
  scales for cognition
Semantic fluency to evaluate neuropsychiatric symptoms | 24 weeks
  scales for language

CONTACTS AND LOCATIONS:
Overall Officials: Sangjin Kim, Professor, Principal Investigator — Inje University Haeundae Paik Hospital
Locations (1):
- Inje university, busan paik hospital, Busan, South Korea

REFERENCES:
- [Background] Ravina B, Putt M, Siderowf A, Farrar JT, Gillespie M, Crawley A, Fernandez HH, Trieschmann MM, Reichwein S, Simuni T. Donepezil for dementia in Parkinson's disease: a randomised, double blind, placebo controlled, crossover study. J Neurol Neurosurg Psychiatry. 2005 Jul;76(7):934-9. doi: 10.1136/jnnp.2004.050682. PMID 15965198
- [Background] Leroi I, Brandt J, Reich SG, Lyketsos CG, Grill S, Thompson R, Marsh L. Randomized placebo-controlled trial of donepezil in cognitive impairment in Parkinson's disease. Int J Geriatr Psychiatry. 2004 Jan;19(1):1-8. doi: 10.1002/gps.993. PMID 14716693
- [Background] Aarsland D, Laake K, Larsen JP, Janvin C. Donepezil for cognitive impairment in Parkinson's disease: a randomised controlled study. J Neurol Neurosurg Psychiatry. 2002 Jun;72(6):708-12. doi: 10.1136/jnnp.72.6.708. PMID 12023410